CLINICAL TRIAL: NCT06531655
Title: Intradetrusor Onabotulinumtoxin A (Botox) at the Time of Transurethral Resection of the Prostate for Mixed Lower Urinary Tract Symptoms
Brief Title: Intradetrusor Botox at the Time of Transurethral Resection of the Prostate for Mixed Lower Urinary Tract Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: TURP procedure bring studied was discontinued due to new Aquablation technology replacing it. Therefore, this study focusing on the outcomes of TURP is being discontinued.
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Cristina Palmer, Principal Investigator, Benaroya Research Institute
Other Study IDs: IRB23-046
Record Dates: First submitted 2024-02-15; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Transurethral Resection of the Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with longstanding obstructive lower urinary tract symptoms (LUTS) due to benign prostatic hypertrophy (BPH) can also develop symptoms of overactive bladder syndrome (OAB). Transurethral resection of the prostate (TURP) is the gold standard treatment for BPH. However, in the immediate post-operative period, TURP can also include OAB-like symptoms, including urinary frequency and urgency. For men with baseline OAB symptoms, this initial worsening of symptoms can be distressing.

Botox is an FDA approved medication with on-label indications to treat overactive bladder. According to AUA guidelines, it is considered a third-line treatment therapy.

The purpose of this study is to evaluate the outcomes of men who have Botox concurrent with their TURP.

DETAILED DESCRIPTION:
An observational study of the effect of Botox injection at the time of TURP will be performed.

If deemed eligible, participants will be invited to participate in this trial. The International Prostate Symptom Score (IPSS) is a questionnaire that is widely used to assess LUTS in patients and assesses for incomplete emptying, frequency, intermittency, urgency, weak stream, hesitancy, and nocturia. The AUA quality of life score (AUA-QoL) asks how these symptoms affect quality of life. When administered as a combined questionnaire, this is referred to as the AUA symptom score. These scores are summed to produce an overall severity score, which can categorize patients as having mild (score 0-7), moderate (8-19) or severe (20-35) LUTS (11). The AUA symptom score is a benchmark in defining the severity of symptoms, and collection of these scores is recommended in the AUA guidelines as part of the initial management of BPH (3,4,12). The UDI-6 is a validated short form of the urogenital distress inventory, and it assesses for the impact and severity of urinary incontinence (13).

Participants will then undergo their TURP and Botox procedure with one of three surgeons in the department of Urology at Virginia Mason.

At approximately four weeks post-op, participants will have a visit with their provider. Symptoms will be assessed by re-administering the AUA symptom score, the UDI-6, PGI-I and the VM Post-Procedure Questionnaire to assess for change in symptoms as well as satisfaction with their procedure.

Participants will then have an approximate 3 month post-op visit, at which time the questionnaires will be re-administered.. Patients will have the opportunity to follow-up with their provider sooner, if needed, based on individual symptoms.

The total expected duration of participation for any given participant is 4 months.

Demographic data, including comorbidities, urodynamics results, post-void residual, uroflow, operative length, estimated blood loss, length of stay, 30 day readmission rate, and 30 day rate of urinary retention will be collected for each subject via the electronic medical record.

We will be evaluating the impact of Botox concurrent with TURP relative to published rates of overactivity and bother after TURP alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age, and being scheduled to undergo TURP and Botox procedure.
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Non-English Speaking
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. History of receiving Botox in the bladder, within the previous 12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include males who have undergone a transurethral resection of the prostate (TURP) as treatment for benign prostatic hypertrophy and obstructive LUTS. The study population will be utilizing Botox as the treatment for overactive bladder (OAB) at the time of TURP.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To identify whether concurrent Botox and TURP are effective at reducing post-operative irritative voiding symptoms. | 1 week
  At the post-operative visit: Trial of Void assessment will be used to assess for rates of postoperative urinary retention.

SECONDARY OUTCOMES:
To identify whether concurrent Botox and TURP lead to higher rates of urinary retention using the American Urological Association symptom score | Four and twelve-week
  Post-op visits when AUA symptom score: (0 to 7 (Mild), 8 to 19 (Moderate), 20 to 35 (Severe))
To identify whether concurrent Botox and TURP lead to rates of urinary retention using internal Virginia Mason Post-Procedure questionnaire | Four and twelve-week
  At the post-operative visit the VM Post Procedure Questionnaire will be administered.
To identify whether concurrent Botox and TURP lead to higher rates of urinary retention using the Patient Global Impression of Improvement (PGI-I) to assess patient observed improvement in urinary incontinence. | Four and twelve-week
  Administer the Patient Global Impression of Improvement (PGI-I)
To identify whether concurrent Botox and TURP lead to higher rates of urinary retention using the Urinary Distress Inventory, Short Form (UDI-6) | Four and twelve-week
  Administer the short 6 question form of the Urinary Distress Inventory at the post-operative visits
To identify whether concurrent Botox and TURP lead to higher rates of urinary retention using a bladder scan to assess the amount of residual urine in bladder post trial of void. | Four and twelve-week
  Post void residual obtained via bladder scan.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Palmer, DO, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng M, Leslie SW, Baradhi KM. Benign Prostatic Hyperplasia. 2024 Oct 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558920/ PMID 32644346
- [Background] Chen LC, Kuo HC. Pathophysiology of refractory overactive bladder. Low Urin Tract Symptoms. 2019 Sep;11(4):177-181. doi: 10.1111/luts.12262. Epub 2019 Mar 22. PMID 30900373
- [Background] Cornu JN, Grise P. Is benign prostatic obstruction surgery indicated for improving overactive bladder symptoms in men with lower urinary tract symptoms? Curr Opin Urol. 2016 Jan;26(1):17-21. doi: 10.1097/MOU.0000000000000249. PMID 26574877
- [Background] Kim SJ, Al Hussein Alawamlh O, Chughtai B, Lee RK. Lower Urinary Tract Symptoms Following Transurethral Resection of Prostate. Curr Urol Rep. 2018 Aug 20;19(10):85. doi: 10.1007/s11934-018-0838-4. PMID 30128964
- [Background] Al-Shaiji TF. Intradetrusor injection of botulinum toxin for the management of refractory overactive bladder syndrome: an update. Surg Innov. 2013 Aug;20(4):351-5. doi: 10.1177/1553350612460125. Epub 2012 Sep 10. PMID 22964263
- [Background] Zillioux J, Welk B, Suskind AM, Gormley EA, Goldman HB. SUFU white paper on overactive bladder anticholinergic medications and dementia risk. Neurourol Urodyn. 2022 Nov;41(8):1928-1933. doi: 10.1002/nau.25037. Epub 2022 Sep 6. PMID 36066046
- [Background] Yap TL, Cromwell DA, Brown C, van der Meulen J, Emberton M. The relationship between objective frequency-volume chart data and the I-PSS in men with lower urinary tract symptoms. Eur Urol. 2007 Sep;52(3):811-8. doi: 10.1016/j.eururo.2007.01.013. Epub 2007 Jan 12. PMID 17276583
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440